CLINICAL TRIAL: NCT01061515
Title: A Phase I Dose-Escalation Trial of Biweekly Intraperitoneal Oxaliplatin With Systemic Capecitabine and Bevacizumab Following Cytoreduction in Patients With Peritoneal Carcinomatosis From Appendiceal or Colorectal Cancer
Brief Title: Biweekly Intraperitoneal Oxaliplatin With Systemic Capecitabine and Bevacizumab for Patients With Peritoneal Carcinomatosis From Appendiceal or Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0136 / 201107017
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma
MeSH Terms: conditions — Carcinoma | interventions — Oxaliplatin; Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose Level 1 (Experimental): Intraperitoneal oxaliplatin 25 mg/m2 IP on day 1 of each cycle
  Bevacizumab 5 mg/kg CIVI on day 1 of each cycle
  Capecitabine PO BID on days 1-7 of each cycle.
  Each cycle is 14 days long.
  Interventions: Drug: Intraperitoneal Oxaliplatin; Drug: Bevacizumab; Drug: Capecitabine
- Dose Level 2 (Experimental): Intraperitoneal oxaliplatin 50 mg/m2 IP on day 1 of each cycle
  Bevacizumab 5 mg/kg CIVI on day 1 of each cycle
  Capecitabine PO BID on days 1-7 of each cycle.
  Each cycle is 14 days long.
  Interventions: Drug: Intraperitoneal Oxaliplatin; Drug: Bevacizumab; Drug: Capecitabine
- Dose Level 3 (Experimental): Intraperitoneal oxaliplatin 65 mg/m2 IP on day 1 of each cycle
  Bevacizumab 5 mg/kg CIVI on day 1 of each cycle
  Capecitabine PO BID on days 1-7 of each cycle.
  Each cycle is 14 days long.
  Interventions: Drug: Intraperitoneal Oxaliplatin; Drug: Bevacizumab; Drug: Capecitabine
- Dose Level 4 (Experimental): Intraperitoneal oxaliplatin 85 mg/m2 IP on day 1 of each cycle
  Bevacizumab 5 mg/kg CIVI on day 1 of each cycle
  Capecitabine PO BID on days 1-7 of each cycle.
  Each cycle is 14 days long.
  Interventions: Drug: Bevacizumab
- Dose Level 5 (Experimental): Intraperitoneal oxaliplatin 100 mg/m2 IP on day 1 of each cycle
  Bevacizumab 5 mg/kg CIVI on day 1 of each cycle
  Capecitabine PO BID on days 1-7 of each cycle.
  Each cycle is 14 days long.
  Interventions: Drug: Intraperitoneal Oxaliplatin; Drug: Bevacizumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Intraperitoneal Oxaliplatin
  Other Names: Eloxatin
  Arms: Dose Level 1; Dose Level 2; Dose Level 3; Dose Level 5
Drug: Bevacizumab
  Other Names: Avastin
Drug: Capecitabine
  Other Names: Xeloda
  Arms: Dose Level 1; Dose Level 2; Dose Level 3; Dose Level 5

SUMMARY:
This study is to test escalating doses of intraperitoneal (IP) oxaliplatin in conjunction with systemic bevacizumab and capecitabine in patients with Peritoneal Carcinomatosis (PC) from either appendiceal or colorectal adenocarcinoma that have been adequately cytoreduced and have undergone a peritoneal scan demonstrating patency of at least one of the intraperitoneal ports that were placed at the time of debulking.

DETAILED DESCRIPTION:
* To determine the maximum tolerated dose of IP oxaliplatin with systemic intravenous bevacizumab and oral capecitabine after adequate surgical debulking and peritoneal scan documenting function of intraperitoneal ports in patients with peritoneal carcinomatosis of appendiceal or colorectal etiology.
* To assess the safety and tolerability of repeated delayed intraperitoneal chemotherapy with oxaliplatin and systemic intravenous bevacizumab and oral capecitabine after adequate surgical debulking and peritoneal scan documenting function of intraperitoneal ports in patients with peritoneal carcinomatosis of appendiceal or colorectal etiology.
* To describe the progression rate, progression-free survival and overall survival in patients treated with this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histological Diagnosis: Patients must have a histologically documented peritoneal carcinomatosis from either colorectal or appendiceal adenocarcinoma.
* Prior Surgical Debulking: Patients must have undergone debulking surgery with peritonectomy and have been allowed at least 4 weeks to recover prior to receiving chemotherapy.
* Port Placement: Intraperitoneal ports may be placed during or at any time separate from surgical debulking. Provided the patient has been allowed at least 4 weeks to recover from surgical debulking, no additional recovery time is required for port placement.
* Active port: Patients must undergo a peritoneal scan documenting at least one working intraperitoneal port prior to receiving chemotherapy.
* Patients may have received prior chemotherapy.
* Age: Patients must be ≥18 years of age. Because no dosing or toxicity data are currently available on the use of oxaliplatin in patients <18 years of age.
* Performance Status: (Eastern cooperativeOncology Group) ECOG 0-2.
* Recovery from Intercurrent Illness: Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmias.
* Informed Consent: All patients must be consented prior to chemotherapy. The patient should not have any serious medical of psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment.
* Hematological Status:

  * absolute neutrophil count ≥1,500/mm³
  * platelet count ≥100,000/mm³
  * hemoglobin ≥8 g/dl.
* Hepatic function:

  * Total bilirubin must be <2X the institutional upper limit of normal (ULN)
  * Transaminases (SGOT and/or SGPT) must be ≤3X the institutional upper limit of normal (ULN)
  * Alkaline phosphatase must be ≤4X the institutional upper limit of normal (ULN)
* Renal Function: Patients must have adequate renal function prior to chemotherapy defined as serum creatinine ≤ 2.0 mg/dl or creatinine clearance ≥60 ml.min/1.73 m² for patients with creatinine levels above 2.0 mg/dl.

Exclusion Criteria:

* Pregnant or breast feeding: For all sexually active patients, the use of adequate contraception (hormonal or barrier method of birth control) will be required during therapy, prior to study entry, and for the duration of study participation. Non-pregnant status will be determined in all women of childbearing potential.
* Prior history of hypersensitivity reactions to oxaliplatin, bevacizumab, 5-FU or capecitabine.
* Gastrointestinal ailments that may alter the absorption of oral medications (i.e. bowel obstruction, short-gut syndrome).
* Patients receiving antiretroviral therapy Highly Active Anti Retroviral Treatment (HAART) for HIV infection are excluded from the study because of possible pharmacokinetic interactions. Appropriate studies will be undertaken in patients receiving HAART therapy, when indicated.
* Patients with Grade 2 or higher peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-05-10 (Actual); Primary Completion 2026-09-27 (Estimated); Study Completion 2026-09-27 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of IP oxaliplatin with systemic intravenous bevacizumab and oral capecitabine after surgical debulking and peritoneal scan documenting functional of intraperitoneal ports in patients with peritoneal carcinomatosis | Completion of enrollment (approximately 8 years)
Assess the safety and tolerability of IP oxaliplatin and intravenous (i.v.) bevacizumab and oral capecitabine after surgical debulking and functional intraperitoneal ports in patients with peritoneal carcinomatosis of appendiceal or colorectal etiology | 30 days after completion of treatment (estimated to be 22 weeks)
Progression rate | Through 4-12 weeks post-treatment (estimated to be 30 weeks)
  -Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-target lesions
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 5 years)
  -Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-target lesions
Overall survival | Through completion of follow-up (estimated to be 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu